CLINICAL TRIAL: NCT04303988
Title: A Prospective, Single-arm, Single-center, Phase II Clinical Study of Triple-negative Breast Cancer Brain Metastases
Brief Title: A Phase II Study of Triple-negative Breast Cancer Brain Metastases.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN 015
Record Dates: First submitted 2020-02-24; First posted 2020-03-11 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort HR-/HER2- (Experimental): Hormone receptor negative, HER2 negative participants will receive SHR1316 in combination with bevacizumab plus cisplatin or carboplatin until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: SHR-1316; Drug: Bevacizumab; Drug: Cisplatin/Carboplatin

INTERVENTIONS:
Drug: SHR-1316 — IV
  Other Names: HTI-1088
Drug: Bevacizumab — IV
  Other Names: Avastin
Drug: Cisplatin/Carboplatin — IV
  Other Names: Bobei

SUMMARY:
Study to assess the effectiveness and safety of SHR 1316, bevacizumab combined with cisplatin/carboplatin for treatment of triple-negative breast cancer brain metastases.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center, Simon's two-stage design, phase II clinical trial in triple-negative breast cancer brain metastases patients. Subjects will receive bevacizumab，SHR1316 combined with cisplatin/carboplatin，and will be treated until disease progression, toxicity is intolerable, informed consent is withdrawn, or investigators determine that medication must be discontinued. Drug efficacy and safety data will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, and ≤ 70 years old, both genders;
2. ECOG performance status 0-2;
3. Pathological tests confirm HR-negative / HER2-negative breast cancer; there is evidence of local recurrence or metastasis；not suitable with curative surgery or radiation therapy；HR negative is defined as: ER-negative and PR-negative, the proportion of positively stained tumor cells in all tumor cells is <1%；HER2- negative is defined as: histologically confirmed to be HER2 IHC (0) or HER2 IHC(1+) or HER2 IHC (2+) and FISH(-);
4. It is required that no platinum drugs have been used before, or platinum drugs have been used (cisplatin/carboplatin only one regimen) and platinum sensitive: no progression during at least 4 cycles of treatment, more than 3 months period between last platinum regimen and the progression of disease；
5. MRI confirmed brain metastases, at least one intracranial parenchymal metastatic lesion with a longest diameter ≥ 1.0 cm without prior radiotherapy；
6. Mannitol or steroid hormone therapy is allowed before enrollment, but the dose of steroid hormone should be stable for at least one week;
7. Adequate function of major organs meets the following requirements:

(1)Blood routine ANC≥1.5×109/L； PLT≥75×109/L； Hb≥90 g/L(Allows blood transfusion or the use of medication to ensure that the content of hemoglobin) (2)Coagulation: INR≤1.5，APTT≤1.5×ULN, PT does not exceed the upper limit of normal (3)Blood biochemistry TBIL≤1.5 × ULN; ALT and AST≤3 × ULN (liver metastasis≤5.0 × ULN); Urea nitrogen ≤ 1.5 × ULN; Cr≤1.5 × ULN or creatinine clearance ≥50 mL / min (Cockcroft-Gault formula) (4)Cardiac ultrasound: LVEF≥50%; (5)12-lead ECG: females QTcF interval <470msec and males <450ms; 8.Willing to join the study, sign informed consent, have good compliance and cooperate with follow-up.

Exclusion Criteria:

1. Leptomeningeal or cystic metastases confirmed by MRI or lumbar puncture.
2. Presence of third interstitial fluid that cannot be controlled by drainage or other methods (e.g., a large amount of pleural effusion and ascites);
3. Whole brain radiotherapy, chemotherapy or surgery within 14 days prior to enrollment. Has received prior therapy with Targeted therapy or Endocrine therapy within the previous week；
4. Subjects with HR-/HER2- who has received prior therapy with bevacizumab or PD-1/PD-L1；
5. Participation in any other clinical trials within 2 weeks of enrollment；
6. Concurrent use of any other Anti-cancer drugs；
7. Other malignancies within 5 years, except cured in-situ of uterine cervix carcinoma , skin basal cell carcinoma and squamous-cell carcinoma；
8. History of heart disease: (1) Arrhythmias requiring medical treatment or clinical significance, (2) Myocardial infarction, (3) Heart failure, (4)Any heart diseases that investigator believes not suitable for this study;
9. History of allergy or hypersensitivity to any of the study drugs or study drug components；
10. History of immunodeficiency including HIV-positive, active hepatitis B/C, other acquired, congenital immunodeficiency disease or history of organ transplantation；
11. A clear history of neurological or mental disorders, including epilepsy or dementia；
12. Pregnant or breastfeeding women. Women of childbearing potential who have a positive pregnancy test or unwilling to use adequate contraception prior to enrollment and for the duration of study participation；
13. According to the investigator's judgment, there is a concomitant disease that seriously endangers the safety of subjects or affects the completion of the study (including but not limited to severe hypertension, severe diabetes, active infection, thyroid disease that cannot be controlled by drugs)；
14. Any condition which in the investigator's opinion makes the subjects unsuitable for the study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate in the CNS | from enrollment to progression or death (for any reason), assessed up to 24 months
  CNS ORR will be assessed by the investigator according to RANO-BM criteria. According to these criteria Complete Response (CR) will be defined as the disappearance of all CNS target lesions sustained for at least 4 weeks; no new lesions, no corticosteroids; stable or improved clinically. Partial Response (PR) will be defined as a decrease of at least 30% in the sum longest diameter (LD) of CNS target lesions, taking as reference the baseline sum LD, sustained for at least 4 weeks; no new lesions; no corticosteroids; stable or improved clinically.

SECONDARY OUTCOMES:
Clinical Benefit Rate in the CNS | from enrollment to progression or death (for any reason), assessed up to 24 months
  CNS clinical benefit rate (CBR) will be defined as the percentage of patients who experience a CR, PR or Stable Disease (SD) for at least 24 weeks.
Progression-free survival | Up to 2 years
  PFS will be defined as the time from the first dose of treatment to death or disease progression.
Overall survival | Up to 2 years
  OS will be defined as the time from the first dose of treatment to death for any cause.
First progression site | Up to 2 years
  The first lesion to progress.
Safety as assessed by percentage of patients with any Adverse Event | Up to 2 years
  Adverse event according to NCI-CTC AE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No